CLINICAL TRIAL: NCT05780177
Title: Brief Behavioral Treatment for Insomnia in Veterans With Posttraumatic Stress Disorder
Acronym: BBTI & PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D4243-R
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder; Insomnia Disorder
Keywords: PTSD; Insomnia
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a randomized, controlled trial of a video- and telephone-based, brief insomnia treatment in Veterans who meet criteria for Insomnia Disorder and Posttraumatic Stress Disorder (PTSD) to accomplish the goal of improving psychosocial functioning.
Who Masked: Outcomes Assessor
Masking Description: The clinical evaluator will be kept blind to treatment condition throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BBTI (Experimental): Participants in this arm will receive 4 sessions (30-60 minutes) of a brief behavioral treatment for insomnia (BBTI). Relaxation techniques are not a component of BBTI.
  Interventions: Behavioral: Brief Behavioral Treatment for Insomnia (BBTI)
- PMRT (Active Comparator): Participants in this arm will receive 4 sessions (30-60 minutes) of progressive muscle relaxation training (PMRT).
  Interventions: Behavioral: Progressive Muscle Relaxation Training (PMRT)

INTERVENTIONS:
Behavioral: Brief Behavioral Treatment for Insomnia (BBTI) — Participants in this arm will receive 4 sessions (30-60 minutes) of a brief behavioral treatment for insomnia called BBTI. Relaxation techniques are not a component of BBTI.
  Arms: BBTI
Behavioral: Progressive Muscle Relaxation Training (PMRT) — Participants in this arm will receive 4 sessions (30-60 minutes) of progressive muscle relaxation training called PMRT.
  Arms: PMRT

SUMMARY:
This study will investigate treatments for insomnia in Veterans who have posttraumatic stress disorder (PTSD). The purpose of this study is to compare a brief behavioral treatment for insomnia (BBTI) to a treatment that helps promote relaxation (progressive muscle relaxation training or PMRT). The investigators will examine improvements in psychosocial functioning and insomnia severity. The investigators will also examine whether treatment gains last over time and whether suicidal ideation decreases following insomnia treatment.

DETAILED DESCRIPTION:
This is a randomized, controlled trial of a video- and telephone-based, brief insomnia treatment in Veterans who meet criteria for Insomnia Disorder and Posttraumatic Stress Disorder (PTSD) to accomplish the goal of improving psychosocial functioning. The primary outcome for the trial will be psychosocial functioning, with insomnia severity serving as the secondary outcome. Additional goals include assessing durability of treatment gains and evaluating whether suicidal ideation decreases after insomnia treatment. Eighty Veterans with Insomnia Disorder and PTSD will be randomly assigned to either Brief Behavioral Treatment for Insomnia (BBTI; one 60-minute and one 45-minute video encounter, and two 30-minute phone-based encounters) or a Progressive Muscle Relaxation Training control group (manualized relaxation training delivered by two video and two phone sessions, matched to the BBTI condition for therapist time). Prior to randomization, participants will complete clinician-administered, mental health diagnostic interviews at baseline (and post-treatment). Self-report measures of psychosocial functioning, insomnia severity, and other mental health symptoms will be completed at baseline (pretreatment), mid-treatment, post-treatment, and at 6-month follow-up (BBTI group only). Sleep parameters will be completed with a self-report sleep diary. One week of sleep parameters data will be collected at baseline and continuously to the post-treatment appointment (and at 6-month follow-up for the BBTI group only). The investigators also will explore whether BBTI decreases suicidal ideation, which often occurs in Veterans with PTSD and insomnia, using the Depressive Symptom Index: Suicidality Subscale and the Columbia Suicide Severity Rating Scale, the latter which is used clinically in VA to assess suicide risk.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-75 years who served in the military
* Veterans who meet DSM-5 Criteria for Insomnia Disorder.
* Veterans who meet DSM-5 Criteria for current PTSD
* If currently taking insomnia, PTSD or other psychotropic medications, must be stable on these medications for at least one month and not make any changes to medications during the active treatment phase of the study.
* If currently receiving any type of psychotherapy, must have received this treatment for at least one month and do not plan to discontinue treatment during the BBTI trial. Individuals planning to start a new type of psychotherapy will be required to wait one month prior to study enrollment. Individuals currently engaged or planning to engage in evidence-based treatments that are recognized by the VA as directly targeting insomnia or PTSD (i.e., Cognitive Behavioral Therapy for Insomnia, Cognitive Processing Therapy, or Prolonged Exposure Therapy) must complete treatment and wait one month prior to screening for the trial.
* The investigators will not exclude individuals with TBI, given that prior studies have found that individuals with mild to severe TBI can benefit from behavioral interventions for insomnia.
* The investigators will not exclude individuals with chronic pain, given that prior studies have found that these individuals can benefit from behavioral interventions for insomnia.
* The investigators will not exclude individuals with treated sleep apnea or untreated sleep apnea or individuals that are high-risk for sleep apnea. Prior research has found that these individuals can benefit from behavioral interventions for insomnia. Recent research has also established that individuals with untreated mild, moderate or severe sleep apnea or those high-risk for sleep apnea are more likely to receive assessment and treatment for this condition after completing behavioral treatment for insomnia.

Exclusion Criteria:

* Veterans with a lifetime history of psychotic disorder or manic episodes.
* Veterans with moderate to severe alcohol or substance use disorder.
* Veterans with recent homicidal behaviors. Veterans with suicidal ideation will not be excluded. However, Veterans with recent suicidal behaviors or hospitalization or those who report prominent suicidal ideation with intent or a plan will be excluded.
* Veterans who are pregnant
* Veterans who work night or rotating shifts
* Veterans with unstable housing
* Veterans with untreated medical conditions that are known to affect sleep (e.g., restless legs syndrome)
* Veterans with uncontrolled seizure disorder. Sleep restriction is contraindicated for people with uncontrolled seizures due to the possibility of triggering a seizure.
* Veterans who are unable to participate in video treatment sessions or complete online surveys.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Work and Social Adjustment Scale (WSAS) Change | Change from baseline (Week 1) to posttreatment (Week 5)
  Assesses functioning in work, home management, social leisure activities, private leisure activities and relationships with others. It is a five-item measure with each item rated on a 0 to 8 scale, with higher scores reflecting greater impairment.
Work and Social Adjustment Scale (WSAS) Change | Change from baseline (Week 1) to 6-month follow-up--for treatment arm only
  Assesses functioning in work, home management, social leisure activities, private leisure activities and relationships with others. It is a five-item measure with each item rated on a 0 to 8 scale, with higher scores reflecting greater impairment.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | Change from baseline (Week 1) to posttreatment (Week 5)
  The ISI is a valid and reliable self-report measure that is a specific index of perceived insomnia severity. The ISI is a 7-item measure that is scored on a five-point Likert scale. Areas assessed include: problems with sleep onset, sleep maintenance, and early morning awakening; dissatisfaction with sleep; interference with daily functioning; impact on quality of life; and worry about sleep problems. Scores of 15 to 21 represent moderate clinical insomnia, and scores of 22 to 28 represent severe clinical insomnia.
Insomnia Severity Index (ISI) | Change from baseline (Week 1) to 6-month follow-up--for treatment arm only
  The ISI is a valid and reliable self-report measure that is a specific index of perceived insomnia severity. The ISI is a 7-item measure that is scored on a five-point Likert scale. Areas assessed include: problems with sleep onset, sleep maintenance, and early morning awakening; dissatisfaction with sleep; interference with daily functioning; impact on quality of life; and worry about sleep problems. Scores of 15 to 21 represent moderate clinical insomnia, and scores of 22 to 28 represent severe clinical insomnia.

OTHER OUTCOMES:
Depressive Symptom Index: Suicidality Subscale (DSI-SS) | Change from baseline (Week 1) to 6-month follow-up--for treatment arm only
  The DSI-SS is a 4-item self-report questionnaire designed to identify the frequency and intensity of suicidal ideation and impulses in the past two weeks. Scores range from 0-12, with higher scores reflecting greater severity of suicidal ideation. The DSI-SS is a reliable and valid measure of severity of SI in psychiatric patients.
Depressive Symptom Index: Suicidality Subscale (DSI-SS) | Change from baseline (Week 1) to posttreatment (Week 5)
  The DSI-SS is a 4-item self-report questionnaire designed to identify the frequency and intensity of suicidal ideation and impulses in the past two weeks. Scores range from 0-12, with higher scores reflecting greater severity of suicidal ideation. The DSI-SS is a reliable and valid measure of severity of SI in psychiatric patients.

CONTACTS AND LOCATIONS:
Overall Officials: Shira Maguen, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No